CLINICAL TRIAL: NCT05332847
Title: Point of Care Ultrasonography Assessment During Pulmonary Hypertension Clinic Changes Patients' Management- A Randomized Controlled Pilot Study
Brief Title: Point of Care Ultrasonography Assessment During Pulmonary Hypertension Clinic
Acronym: POCUSPAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Avital Keren Abriel MD, Head of Pulmonary Hypertension clinic, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 032716SOR
Record Dates: First submitted 2022-03-13; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: POCUS Assessment During Ambulatory PAH Clinic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The intervention group underwent clinical evaluation and a bedside-focused sonographic assessment
  Interventions: Device: POC-US
- control group. (No Intervention): The control group underwent clinical evaluation without POC-US

INTERVENTIONS:
Device: POC-US — Point Of Care Ultrasonography (POCUS) is a rapidly evolving bedside modality in which ultrasonography is utilized as a part of the bedside physical examination and the patients' clinical assessment
  Other Names: clinic visit evaluations
  Arms: intervention group

SUMMARY:
Background: Changes occurring in the pulmonary vascularity imparts changes to the right heart in patients with pulmonary arterial hypertension (PAH). Importantly changes in RV function correlates with severity of disease and patient outcome. This affords and opportunity to assess patients longitudinally through point of care ultrasonography. Investigators objective was to measure the percentage and the rate of patients management change, represented by change in treatment or assessment of patients in the PAH clinic, and to compared management change rate between patients with PAH who underwent point of care ultrasonography (POCUS) assessment in addition to the routine evaluation, and a control group to which the investigators did not add a test with POCUS in addition to the routine evaluation in the clinic.

Methods: Consecutive patients from the PAH clinic in two medical centers were randomized to the POCUS assessment group and the non-POCUS group. The POCUS group received lung, heart, and vascular ultrasound assessments. All other assessments were the same between both groups. Management changes were documented during each of the patients' visits over a three-month interval.

DETAILED DESCRIPTION:
The investigators included patients if they were diagnosed with group 1 PH (PAH), as defined by the updated clinical classiﬁcation of PH and provided informed consent. Patients were excluded if diagnosed with PH group 2-5, had congenital heart disease, liver cirrhosis, or suspected pulmonary venous-occlusive disease. On enrollment, randomization of the patient was done 1:1 (using ClinStat) to either the POCUS assessment group or control group. Both groups underwent the same clinical assessment according to PH clinic protocol and by the same treating pulmonologist (A.A.). Every patient was scheduled to a follow up meeting every three months as part of the usual PAH clinic routine. The study protocol was approved by each participating center's research ethics board (BRZ 0106-18, SOR0327-16).

At each clinic visit evaluations for both groups were standardized. Each visit included a history, physical and laboratory evaluation, BNP level, 6-minute walk test, and quality of life as assessed using emPHasis 10.

Prior to the decision regarding patient management, the pulmonologist at the PAH clinic knew the test results including a POCUS test done in the intervention group. A change in the patient's management in the clinic is represented by the clinician's recommendation for a change in medication, sending the patient for a lung transplant, hospitalization, or other diagnostic or therapeutic procedure documented

Patients in the intervention group underwent a bedside-focused sonographic assessment of the heart, lungs, abdomen, and IVC in every clinic visit during the period of study. The exam was conducted either at the beginning or after the regular patient assessment. The Investigators used 2-dimensional views, the parasternal long and short axis, subcostal long and IVC, apical 5, 4, 2 chamber view. As this exam was POCUS centered and not a formal cardiac study. When pathologies were identified, relevant measurements were made, and the patient was referred for a formal echo. For example, when a calcified aortic valve was detected, and aortic stenosis was suspected a continuous pulse wave Doppler for maximal velocity measurement was conducted. Standard measurements were for left ventricle wall thickness, size of ventricles and atria, IVC size and collapsibility index, RVSP when TR was identified, TAPSE, and size of pericardial effusion when found. Lung ultrasound was focused on the detection of pulmonary congestion (screening and counting B-lines on both lungs, midclavicular line and midaxillary line), pleural effusion, lung atelectasis, lung consolidations (mid and posterior axillary lines), and sliding of pleura (midclavicular line). The investigators performed Doppler for DVT only within the right clinical context. All POCUS exams were documented in a standardized form. Findings were reported in real-time to the treating pulmonologist and were documented in the follow-up notes.

ELIGIBILITY:
Inclusion Criteria:

* All patients with PAH defined by the Updated clinical classiﬁcation of pulmonary hypertension criteria.
* Age ≥ 18
* Baseline values from right-heart catheterization results for the definite diagnosis of PH: Hemodynamic inclusion: resting mPAP > 25mmHg, PCWP < 15mmHg, and PVR > 3 Woods Units.

Exclusion Criteria:

* Inability to give informed consent.
* Clear evidence of Group 2-5 PH. We will also exclude patients with PAH on the basis of congenital heart disease, liver cirrhosis or suspected pulmonary veno-occlusive disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-01-14 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
percentage and the rate of patients management change, represented by change in treatment or assessment of patients in the PAH clinic | 9 monthes

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Medical Center, Beersheba, Negev, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Avriel A, Bar Lavie Shay A, Hershko Klement A, Taylor J, Shamia D, Tsaban G, Abu-Shakra M, Granton J, Fuchs L. Point-of-Care Ultrasonography in a Pulmonary Hypertension Clinic: A Randomized Pilot Study. J Clin Med. 2023 Feb 22;12(5):1752. doi: 10.3390/jcm12051752. PMID 36902536